CLINICAL TRIAL: NCT00005520
Title: Genetic Epidemiology of Responses to Antihypertensives
Acronym: GERA
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen T. Turner, Professor of Medicine, Mayo Clinic
Other Study IDs: 05-004017; R01HL053330 (NIH); R01HL074735 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
Keywords: Hypertension; Pharmacogenetics; Hydrochlorothiazide; Candesartan
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Hydrochlorothiazide; candesartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- African American hydrochlorothiazide: 300 African American hypertensives were treated with hydrochlorothiazide 25 mg daily for 4 weeks.
  Interventions: Drug: Hydrochlorothiazide
- European American hydrochlorothiazide: 300 European American hypertensives were treated with hydrochlorothiazide 25 mg daily for 4 weeks
  Interventions: Drug: Hydrochlorothiazide
- African American candesartan: 300 African American hypertensives were treated with candesartan 16 mg daily for 2 weeks followed by 32 mg daily for 4 weeks
  Interventions: Drug: Candesartan
- European American candesartan: 300 European American hypertensives were treated with candesartan 16 mg daily for 2 weeks followed by 32 mg daily for 4 weeks
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Hydrochlorothiazide
  Groups: African American hydrochlorothiazide; European American hydrochlorothiazide
Drug: Candesartan
  Groups: African American candesartan; European American candesartan

SUMMARY:
To determine whether measured variation in genes coding for components of vasoconstriction and volume regulating systems predict interindividual differences in blood pressure response to therapy with a thiazide diuretic, hydrochlorothiazide, or an angiotensin II receptor blocker, candesartan, in hypertensive African-Americans (N=300 treated with each drug) and in hypertensive European Americans (N=300 treated with each drug).

DETAILED DESCRIPTION:
BACKGROUND:

Essential hypertension is a common disorder that contributes to morbidity, mortality, and cost of health care, especially among African-Americans. Although a single-drug therapy is commonly prescribed for treatment of hypertension, blood pressure levels are controlled in some individuals but not in others. The study has the potential to identify genes contributing to the etiology of interindividual differences in blood pressure response to diuretic therapy in African-Americans and European Americans.

DESIGN NARRATIVE:

Hypertensive adults were treated with the diuretic hydrochlorothiazide, 25 mg/day, for four weeks; or with the angiotensin II receptor blocker candesartan, 16 mg/day for 2 weeks followed by 32 mg/day for 4 weeks. Interindividual variations in blood pressure responses and in candidate genes coding for components of systems regulating vasoconstriction and volume were measured. In addition, a panel of 500,000 single nucleotide polymorphisms genome-wide was measured in subsets of the most extreme responders and nonresponders to each drug for genome-wide association of analyses.

ELIGIBILITY:
Primary (essential) hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult African American men and women with previously diagnosed primary hypertension were recruited from Atlanta, Georgia; and adult European American man and women with previously diagnosed primary hypertension were recruited from Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 1997-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 4 weeks for hydrochlorothiazide; 6 weeks for candesartan
  The blood pressure response to antihypertensive drug therapy was defined by the difference between blood pressure levels prior to and at the end of drug therapy.

SECONDARY OUTCOMES:
Adverse metabolic changes | 4 weeks for hydrochlorothiazide only
  Potentially adverse metabolic changes in response to hydrochlorothiazide include changes in fasting serum glucose and insulin; serum potassium; serum lipids (triglycerides, HDL-cholesterol, total cholesterol); and serum uric acid.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T. Turner, M.D., Principal Investigator — Mayo Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Turner ST, Schwartz GL, Chapman AB, Boerwinkle E. C825T polymorphism of the G protein beta(3)-subunit and antihypertensive response to a thiazide diuretic. Hypertension. 2001 Feb;37(2 Pt 2):739-43. doi: 10.1161/01.hyp.37.2.739. PMID 11230366
- [Background] Turner ST, Boerwinkle E. Genetics of hypertension, target-organ complications, and response to therapy. Circulation. 2000 Nov 14;102(20 Suppl 4):IV40-5. doi: 10.1161/01.cir.102.suppl_4.iv-40. No abstract available. PMID 11080130
- [Background] Turner ST, Schwartz GL, Chapman AB, Hall WD, Boerwinkle E. Antihypertensive pharmacogenetics: getting the right drug into the right patient. J Hypertens. 2001 Jan;19(1):1-11. doi: 10.1097/00004872-200101000-00001. PMID 11204288
- [Background] Montori VM, Schwartz GL, Chapman AB, Boerwinkle E, Turner ST. Validity of the aldosterone-renin ratio used to screen for primary aldosteronism. Mayo Clin Proc. 2001 Sep;76(9):877-82. doi: 10.4065/76.9.877. PMID 11560297
- [Background] Turner ST, Schwartz GL, Chapman AB, Boerwinkle E. Use of gene markers to guide antihypertensive therapy. Curr Hypertens Rep. 2001 Oct;3(5):410-5. doi: 10.1007/s11906-001-0059-x. PMID 11551376
- [Background] Schwartz GL, Chapman AB, Boerwinkle E, Kisabeth RM, Turner ST. Screening for primary aldosteronism: implications of an increased plasma aldosterone/renin ratio. Clin Chem. 2002 Nov;48(11):1919-23. PMID 12406976
- [Background] Garovic VD, Joyner MJ, Dietz NM, Boerwinkle E, Turner ST. Beta(2)-adrenergic receptor polymorphism and nitric oxide-dependent forearm blood flow responses to isoproterenol in humans. J Physiol. 2003 Jan 15;546(Pt 2):583-9. doi: 10.1113/jphysiol.2002.031138. PMID 12527744
- [Background] Turner ST, Boerwinkle E. Genetics of blood pressure, hypertensive complications, and antihypertensive drug responses. Pharmacogenomics. 2003 Jan;4(1):53-65. doi: 10.1517/phgs.4.1.53.22587. PMID 12517286
- [Background] Schwartz GL, Turner ST. Pharmacogenetics of antihypertensive drug responses. Am J Pharmacogenomics. 2004;4(3):151-60. doi: 10.2165/00129785-200404030-00002. PMID 15174896
- [Background] Frazier L, Turner ST, Schwartz GL, Chapman AB, Boerwinkle E. Multilocus effects of the renin-angiotensin-aldosterone system genes on blood pressure response to a thiazide diuretic. Pharmacogenomics J. 2004;4(1):17-23. doi: 10.1038/sj.tpj.6500215. PMID 14735111
- [Background] Turner ST, Chapman AB, Schwartz GL, Boerwinkle E. Effects of endothelial nitric oxide synthase, alpha-adducin, and other candidate gene polymorphisms on blood pressure response to hydrochlorothiazide. Am J Hypertens. 2003 Oct;16(10):834-9. doi: 10.1016/s0895-7061(03)01011-2. PMID 14553962
- [Background] Finkielman JD, Schwartz GL, Chapman AB, Boerwinkle E, Turner ST. Lack of agreement between office and ambulatory blood pressure responses to hydrochlorothiazide. Am J Hypertens. 2005 Mar;18(3):398-402. doi: 10.1016/j.amjhyper.2004.10.021. PMID 15797660
- [Background] Turner ST, Schwartz GL. Gene markers and antihypertensive therapy. Curr Hypertens Rep. 2005 Feb;7(1):21-30. doi: 10.1007/s11906-005-0051-y. PMID 15683583
- [Background] Schwartz GL, Turner ST. Screening for primary aldosteronism in essential hypertension: diagnostic accuracy of the ratio of plasma aldosterone concentration to plasma renin activity. Clin Chem. 2005 Feb;51(2):386-94. doi: 10.1373/clinchem.2004.041780. PMID 15681560
- [Background] Maitland-van der Zee AH, Turner ST, Schwartz GL, Chapman AB, Klungel OH, Boerwinkle E. A multilocus approach to the antihypertensive pharmacogenetics of hydrochlorothiazide. Pharmacogenet Genomics. 2005 May;15(5):287-93. doi: 10.1097/01213011-200505000-00003. PMID 15864129
- [Result] Turner ST, Schwartz GL, Chapman AB, Beitelshees AL, Gums JG, Cooper-Dehoff RM, Boerwinkle E, Johnson JA, Bailey KR. Power to identify a genetic predictor of antihypertensive drug response using different methods to measure blood pressure response. J Transl Med. 2012 Mar 13;10:47. doi: 10.1186/1479-5876-10-47. PMID 22413836
- [Derived] Chekka LMS, Tantawy M, Langaee T, Wang D, Renne R, Chapman AB, Gums JG, Boerwinkle E, Cooper-DeHoff RM, Johnson JA. Circulating microRNA Biomarkers of Thiazide Response in Hypertension. J Am Heart Assoc. 2024 Feb 20;13(4):e032433. doi: 10.1161/JAHA.123.032433. Epub 2024 Feb 14. PMID 38353215
- [Derived] Mehanna M, Wang Z, Gong Y, McDonough CW, Beitelshees AL, Gums JG, Chapman AB, Schwartz GL, Bailey KR, Johnson JA, Turner ST, Cooper-DeHoff RM. Plasma Renin Activity Is a Predictive Biomarker of Blood Pressure Response in European but not in African Americans With Uncomplicated Hypertension. Am J Hypertens. 2019 Jun 11;32(7):668-675. doi: 10.1093/ajh/hpz022. PMID 30753254
- [Derived] Duarte JD, Zineh I, Burkley B, Gong Y, Langaee TY, Turner ST, Chapman AB, Boerwinkle E, Gums JG, Cooper-Dehoff RM, Beitelshees AL, Bailey KR, Fillingim RB, Kone BC, Johnson JA. Effects of genetic variation in H3K79 methylation regulatory genes on clinical blood pressure and blood pressure response to hydrochlorothiazide. J Transl Med. 2012 Mar 22;10:56. doi: 10.1186/1479-5876-10-56. PMID 22440088